CLINICAL TRIAL: NCT02950077
Title: Mindfulness - Based Stress Reduction and the Relationship on Inflammation in Autoimmune Hepatitis - A Human Pilot Study Protocol
Brief Title: Mindfulness - Based Stress Reduction and the Relationship on Inflammation in Autoimmune Hepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000020043
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Individuals who are under the care of the Yale Liver Center with a diagnosis of autoimmune hepatitis
  Interventions: Behavioral: mindfulness based stress reduction

INTERVENTIONS:
Behavioral: mindfulness based stress reduction — The intervention will be delivered in a group setting and the group will meet for 2 hours once per week for 8 weeks. The intervention is based on new neuroscience of stress and resilient adaptive behaviors, mindfulness based stress reduction, therapeutic breath and synchronized yogic movement with a focus on the lower abdomen, integrated with cognitive and behavioral strategies for self-control and healthy decision making.

SUMMARY:
The study is a 'pilot study' to assess the effect of a mindfulness-based stress reduction (MBSR) intervention on patients with autoimmune liver disease specifically autoimmune hepatitis type I. MBSR is a standardized intervention that has shown benefit in addiction disorders and other psychiatric disorders. There has been no study evaluating or showing the benefit of the use of MBSR in autoimmune liver disease. With published data showing the evidence of an association of stress and relapse in autoimmune hepatitis, it is hypothesized that such an intervention such as MBSR may have therapeutic effect in patients with autoimmune liver disease.

DETAILED DESCRIPTION:
With the understanding that autoimmune hepatitis has a relationship with psychological stress, the use of a strategy such as mindfulness stress based reduction (MBSR) may similarly have a substantial impact as seen in other disease conditions. The proposed hypothesis is that undergoing MBSR has potential to benefit patients with autoimmune hepatitis in relation to decreased relapse rate and ultimately improved quality of life.

The focus of this study is surrounding the possibility of psychosocial stress for relapse in AIH. The investigators, however, would like to also understand the role of serological testing at the time of these relapses and during states of psychosocial stress to demonstrate if the association can be found. During active disease activity or relapses of autoimmune hepatitis, there is an expected rise in alanine aminotransferase (ALT) and immunoglobulin G (IgG) levels. Demonstrating the correlation of ALT and IgG with disease status and possible improvement with stress modifications is also key for this proposed study.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18-80 years
* Diagnosis of Autoimmune Hepatitis Type I

Exclusion Criteria:

Medical

* Hospitalization in the last 30 days
* New immunosuppression agent started <6 weeks prior to study
* Patients with concurrent viral hepatitis and/or alcoholic liver disease
* Patients with decompensated cirrhosis (defined as ascites, encephalopathy, variceal hemorrhage)
* Patients with hepatocellular carcinoma
* Patients post-liver transplantation Psychological
* Any psychotic disorder or current psychiatric symptoms

Attitudinal

* Inability to commit to program schedule and attendance of classes

Physical

* Inability to physically attend classes; disability or physical impairment not included as an exclusion criteria Other
* Inadequate English proficiency
* Inability to read and/or write

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Change in Subjective Stress: The Perceived Stress Scale | 12 months
  Subjective Stress: The Perceived Stress Scale, a 14-item self-report scale that assesses the degree to which individuals appraise situations in their lives as stressful, will be used to assess subjective interpretation of stress and assign subjects to the low stress or high stress condition. Scale It has excellent test-retest reliability and good construct validity and has been used with adults and adolescents.
  Scale ranges from 0 to 40. A higher score indicates higher stress.
Change in Recent Life Stress: Life Experience Survey | 12 months
  The LES is a widely used 57 item self-report measure. It shows convergent validity with personality measures (e.g., anxiety) and is not correlated with social desirability measures.
  Scale ranges from -250 to +250. A higher score indicates higher stress.
Daily Hassles Questionnaire | 12 months
  This self-report item measures how stressful subjects perceived situations occurring in the past year of their life.
  Scale ranges from 0 to 351. A higher score indicates higher stress.
The Brief Self-Control Scale | 12 months
  The Brief Self-Control Scale will be used to measure self-reported self-control and impulsivity. The BSCS also shows good internal consistency (alphas = .83 - .84) and high retest reliability (.87).
  Scale ranges from 13-65. A higher score indicates better self-control.

SECONDARY OUTCOMES:
Change in ALT levels and IgG levels | 12 months
  Abnormal AST and ALT will be defined as >2x upper limits of normal
  Normal Lab ranges that will be used are the following:
  * AST (0 - 34 U/L)
  * ALT (0 - 34 U/L)
  * IgG (355 - 1887 mg/dL)
  These levels are used together for clinical significance and diagnosis.
Change in average medication needed | 12 months
  E.g (changes in monthly prednisone dose)
Change in number of relapses | up to 2 years
  Relapse is defined in one of two ways once immunosuppression has been tapered off:
  I. An increase in the AST or ALT ≥2 X ULN (upper limit of normal) II. An increase in AST and/or ALT ≥ 2 X the prior level of AST or ALT on routine labs checked at start of clinical study
Demonstration of MIF and CD74 have a role as a biomarker for disease activity | 12 months
  Demonstration of a correlation of serum MIF and CD74 levels with autoimmune hepatitis disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: James Boyer, MD, Principal Investigator — Yale University; David Assis, MD, Study Director — Yale University
Locations (1):
- Yale Liver Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alrabadi LS, Dutton A, Rabiee A, Roberts SJ, Deng Y, Cusack L, Silveira MG, Ciarleglio M, Bucala R, Sinha R, Boyer JL, Assis DN. Mindfulness-based stress reduction may decrease stress, disease activity, and inflammatory cytokine levels in patients with autoimmune hepatitis. JHEP Rep. 2022 Feb 18;4(5):100450. doi: 10.1016/j.jhepr.2022.100450. eCollection 2022 May. PMID 35434588